CLINICAL TRIAL: NCT00466843
Title: Mechanism and Response of Thymoglobulin in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Effects of Antithymocyte Globulin in Adults With Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Office of Rare Diseases (ORD) (NIH)
Collaborators: Rare Diseases Clinical Research Network (Network)
Responsible Party: Alan List, MD, H. Lee Moffitt Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDCRN 5406
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Abnormal hematopoiesis; Leukemia; Autoimmune Disease
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Autoimmune Diseases | interventions — Antilymphocyte Serum; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will be treated with ATG
  Interventions: Drug: Antithymocyte globulin (ATG); Drug: Prednisone

INTERVENTIONS:
Drug: Antithymocyte globulin (ATG) — ATG 2.5 mg/kg/day via IV will be given for 4 doses. Each participant will receive only one cycle of therapy. The daily infusion will be administered over at least 6 hours and slowed as necessary to minimize infusion-related symptoms.
Drug: Prednisone — All participants will be pre-treated with prednisone (1 mg/kg/day by mouth) 2 days prior to the first ATG does and continuing for 14 days after the final dose to prevent serum sickness

SUMMARY:
Myelodysplastic syndrome (MDS) is a rare, potentially serious bone marrow disease. Currently available treatments for MDS have been only somewhat beneficial. The purpose of this study is to determine the effects of the medication antithymocyte globulin (ATG) in adults with MDS and to determine which individuals with MDS are most likely to benefit from treatment with ATG.

DETAILED DESCRIPTION:
In people with MDS, the bone marrow stops making healthy blood cells and instead produces poorly functioning, malformed, and immature blood cells. This can lead to anemia resulting from too few healthy red blood cells, infection resulting from too few healthy white blood cells, and bleeding resulting from too few healthy platelets. The exact cause of MDS remains unknown, but it may be caused by abnormal autoimmune activity in which activated T cells, a type of white blood cell, prevent normal bone marrow production. ATG, a medication that inhibits immune function, can restore normal blood production in some people with MDS, but it is not known how this happens and why it does not happen in all MDS patients. The purpose of this study is to examine the effects of ATG in adults with MDS and to determine which individuals with MDS are most likely to benefit from treatment with ATG.

Based on disease severity and likely disease progression, participants will be separated into either a high-risk group or a low-risk group. Participants will be hospitalized for a 4-day period during which they will receive daily infusions of ATG. Oral prednisone will be given 2 days before hospitalization, throughout hospitalization, and then for 14 days after hospitalization to limit the side effects of ATG. Antihistamines and acetaminophen will also be given during hospitalization to reduce the chances of an allergic reaction to ATG. After discharge, all participants will attend monthly study visits that will include blood collection, review of disease symptoms, and evaluation of medication response. At Week 16, participants in the high-risk group will undergo additional blood collection, a bone marrow biopsy, and a thorough evaluation of disease progression and the effects of MDS on daily living abilities. Participants in the low-risk group will undergo these same procedures at Week 24. Follow-up for all participants may last up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS that meets International Prognostic Scoring System (IPSS) criteria for low risk, intermediate-1 risk, or intermediate-2 risk. More information about this criterion can be found in the protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Willing and able to attend study visits
* Willing to use acceptable forms of contraception prior to study entry and for the duration of the study

Exclusion Criteria:

* Any serious medical illness that might limit survival to less than 2 years
* Any other uncontrolled condition or illness. More information about this criterion can be found in the protocol.
* Prior anti-lymphocyte serotherapy (received serum from an immunized animal)
* Proliferative chronic myelomonocytic leukemia
* MDS that is caused by radiotherapy, chemotherapy, and/or immunotherapy for cancerous or autoimmune diseases
* Previous or current cancer. More information about this criterion can be found in the protocol.
* Receiving any other investigational agents
* Certain abnormal lab values. More information about this criterion can be found in the protocol.
* History of a grade 2 National Cancer Institute common toxic criteria allergic reaction to rabbit proteins
* Psychiatric illness that might interfere with study participation
* HIV-1 infection
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Bone marrow response and hematologic improvement | Measured at Week 16 or 24
Bone marrow cytogenetic response | Measured at Week 16 or 24

CONTACTS AND LOCATIONS:
Overall Officials: Alan List, MD, Principal Investigator — H. Lee Moffitt Cancer Center
Locations (4):
- United States (4):
  - UCLA Oncology Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic Foundation - Case Western University, Cleveland, Ohio
  - Penn State University, Hershey, Pennsylvania

REFERENCES:
- [Background] Kochenderfer JN, Kobayashi S, Wieder ED, Su C, Molldrem JJ. Loss of T-lymphocyte clonal dominance in patients with myelodysplastic syndrome responsive to immunosuppression. Blood. 2002 Nov 15;100(10):3639-45. doi: 10.1182/blood-2002-01-0155. Epub 2002 Jul 5. PMID 12393644
- [Background] Maciejewski JP, Rivera C, Kook H, Dunn D, Young NS. Relationship between bone marrow failure syndromes and the presence of glycophosphatidyl inositol-anchored protein-deficient clones. Br J Haematol. 2001 Dec;115(4):1015-22. doi: 10.1046/j.1365-2141.2001.03191.x. PMID 11843844
- [Background] Molldrem JJ, Leifer E, Bahceci E, Saunthararajah Y, Rivera M, Dunbar C, Liu J, Nakamura R, Young NS, Barrett AJ. Antithymocyte globulin for treatment of the bone marrow failure associated with myelodysplastic syndromes. Ann Intern Med. 2002 Aug 6;137(3):156-63. doi: 10.7326/0003-4819-137-3-200208060-00007. PMID 12160363
- [Derived] Komrokji RS, Mailloux AW, Chen DT, Sekeres MA, Paquette R, Fulp WJ, Sugimori C, Paleveda-Pena J, Maciejewski JP, List AF, Epling-Burnette PK. A phase II multicenter rabbit anti-thymocyte globulin trial in patients with myelodysplastic syndromes identifying a novel model for response prediction. Haematologica. 2014 Jul;99(7):1176-83. doi: 10.3324/haematol.2012.083345. Epub 2014 Jan 31. PMID 24488560